CLINICAL TRIAL: NCT02297945
Title: Prospective, Single Arm, Open-label, Multicenter, International Study to Assess the Effects of Metyrapone in Patients With Endogenous Cushing's Syndrome During a 12-week Treatment Period Followed by an Extension Period of 24 Weeks
Brief Title: Effects of Metyrapone in Patients With Endogenous Cushing's Syndrome
Acronym: PROMPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRA112025-002
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cushing's Syndrome
MeSH Terms: conditions — Cushing Syndrome | interventions — Metyrapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metyrapone (Experimental): Metyrapone will be administered orally in an open-label fashion. Two possible initiation doses will be used depending on the severity of hypercortisolism, dose will then be adjusted (up or down-titrated) during the first month on an individual basis according to clinical tolerance and cortisol levels achieved.
  Interventions: Drug: metyrapone

INTERVENTIONS:
Drug: metyrapone — Single arm study
  Other Names: Metopirone

SUMMARY:
The purpose of this prospective, international phase III/IV study is to assess the efficacy and safety of metyrapone in patients with endogenous Cushing's syndrome during up to 36 weeks of treatment. The ability of metyrapone (250 mg capsules) to normalize urinary free cortisol (UFC) levels will be assessed during up to 36 weeks (9 months) of treatment.

DETAILED DESCRIPTION:
This study will include Cushing disease patients with persistent or recurrent disease (after pituitary surgery) or who are newly diagnosed but are unsuitable for early surgery or wish to defer surgery. It will also include patients with ectopic ACTH syndrome (either occult, after surgery failure, or inoperable or metastatic) and patients with Cushing's syndrome from adrenal causes.

The ability of metyrapone to normalize urinary free cortisol levels will be assessed during up to 36 weeks (9 months) of treatment. Patients participating in this study and who are controlled or close to the target at the end of a 3-months period may continue with an optional extension period of 6 months in which the long-term efficacy and safety profiles of metyrapone will be assessed. This extension study is intended to provide new findings to consolidate existing efficacy and safety data on metyrapone in the treatment of Cushing's syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with endogenous Cushing's syndrome:

* Cushing disease patients with persistent or recurrent disease (after pituitary surgery) or who are newly diagnosed but are unsuitable for early surgery or wish to defer surgery;
* Patients with ectopic ACTH syndrome (either occult, after surgery failure, or inoperable or metastatic);
* Patients with Cushing's syndrome from adrenal causes

Exclusion Criteria:

1. Pseudo Cushing's syndrome
2. Cyclic Cushing's syndrome defined by at least one normal UFC value among at least three 24-hour urinary sampling measurements over the previous 2 months
3. Advanced adrenocortical carcinoma or ectopic ACTH secretion (EAS) secondary to a small cell lung carcinoma
4. Life expectancy less than 3 months
5. Pituitary or adrenal surgery or pituitary irradiation or surgery of the ACTH-secreting ectopic tumor or bilateral adrenalectomy planned before the week 12 visit
6. Pituitary irradiation within the previous 5 years (for Cushing's disease patients)
7. Enlarged pituitary adenoma (greater than 1 cm in vertical diameter and leaving less than 2 mm from the chiasma) or compression of the optic chiasma on the pituitary MRI for patients with Cushing's disease
8. Severe uncontrolled hypertension (>180/110 mmHg) despite anti-hypertensive therapy (for otherwise eligible patients, blood pressure medication may be adjusted to meet this criterion)
9. Severe hypokalemia (< 2.5 mmol/L) despite corrective measures
10. White blood cell counts <3 x 109 /L; hemoglobin <10 g/dL; platelets <100 x 109 /L
11. Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that in the judgment of the investigator, would present excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Normalization of cortisol levels (urinary free cortisol) | 3 months

CONTACTS AND LOCATIONS:
Locations (36):
- Belgium (4):
  - University hospital Antwerp, Antwerp
  - CHU Erasme, Brussels
  - University hospital Saint Luc, Brussels
  - CHU Liège, Liège
- Germany (4):
  - Charité Berlin, Berlin
  - Universitätsklinikum Essen, Essen
  - Munich university, Munich
  - University hospital Wuerzburg, Würzburg
- Hungary (5):
  - State health center, Budapest
  - Semmelweis Egyetem II. Belgyógyászati Klinika, Budapest
  - University Debrecen, Debrecen
  - University of Pecs, Pécs
  - University of Szeged, Szeged
- Italy (7):
  - San Luigi Gonzaga Hospital, University of Turin, Orbassano, Turin
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Luca IRCCS Istituto Auxologico Italiano, Milan
  - S. Giuseppe Hospital, Milan
  - Federico II University, Naples
  - University of Padova, Padua
  - University of Turin, Turin
- Poland (3):
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice
  - University Hospital, Krakow
  - University Clinical Hospital, Wroclaw
- Romania (7):
  - Institutul National de Endocrinologie 'C.I Parhon' - Endocrinologie II, Bucharest
  - Institutul National de Endocrinologie 'C.I Parhon' - Endocrinologie VI, Bucharest
  - Spitalul Universitar de Urgenta Militar Central 'Dr Carol Davila', Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - S.C Centrul Clinic Mediquest SRL, Sângeorgiu de Mureş
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- Spain (2):
  - University hospital clinic of Barcelona, Barcelona
  - Hospital Universitario La Ribera, Valencia
- Turkey (Türkiye) (4):
  - Ankara Numune Training and Research Hospital, Ankara
  - Dokuz Eylul UMF, Izmir
  - Ondokuz Mayıs University Medical Faculty, Samsun
  - Karadeniz Teknik University, Trabzon